CLINICAL TRIAL: NCT02297581
Title: A Prospective Multicenter Cohort Study to Evaluate the Benefit of the Geriatric Fracture Center (GFC) Concept
Brief Title: Geriatric Fracture Centers - Evaluation of a Geriatric Co-management Program
Status: Completed | Type: Observational
Sponsor: AO Innovation Translation Center (Other)
Responsible Party: Sponsor
Other Study IDs: GFC
Record Dates: First submitted 2014-11-17; First posted 2014-11-21 (Estimated); Last update posted 2020-06-04 (Actual); Status verified 2019-01

CONDITIONS: Hip Fractures
Keywords: Geriatrics [MeSH]; Osteoporotic fractures [MeSH]; Hip fractures [MeSH]; Cost benefit analysis [MeSH]; Quality of life [MeSH]; Mortality [MeSH]; Complications
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- GFC: Geriatric Fracture Center: Patient treatment in a geriatric fracture center
  A GFC is defined as follows:
  * General geriatrician or ortho-geriatrician available in trauma/orthopaedic department
  * Geriatrician sees the patient prior to surgery (except if the patient is admitted over night or during weekends)
  * Local medical guidelines, consented by orthopedic surgeons and geriatrician
  * Pre-defined order set for assessing laboratory values
  * Pre-defined patient pathway to guarantee a fast track in the emergency room
  * Daily communication among involved specialists
  * Postoperative phase up to discharge from orthopaedic / trauma department (i.e. Discharge 1):
    * Daily patient visit by geriatrician
    * Daily patient visit by orthopedic surgeon in combination with nurse
    * Daily therapy by physiotherapists, except for weekends
    * Access to social workers, if required
- UCC: Usual Care Center: Patient treatment in an usual care center
  A UCC is defined as follows:
  * No geriatrician available in trauma/orthopaedic department
  * No pre-operative visit by a geriatrician as a standard
  * No pre-defined medical guidelines for geriatric fracture patients
  * Postoperative phase up to discharge from orthopaedic / trauma department (i.e. Discharge 1):
    * No daily patient visits by a geriatrician as a standard

SUMMARY:
The study will assess patients with at least one major AE related to treatment / hospitalization / immobilization in the Geriatric Fracture Center (GFC) group compared to the usual care group.

DETAILED DESCRIPTION:
Patients aged ≥ 70 years or older with an osteoporotic hip fracture treated with an osteosynthesis or endoprosthesis will be included in this study.

The primary objective of the study is to assess the difference in the numbers of pre-defined major adverse events (AE) which are related to the treatment, hospitalization and/or immobilization between patients who were treated in a geriatric fracture center or in a usual care center.

As a secondary objective, health economic implications and cost-effectiveness comparison analyses will be performed.

In order to be able to analyze data based on the geographic regions as well as globally, in each participating country, both a Geriatric Fracture Center (GFC) and a Usual Care Center (UCC) will be included.

ELIGIBILITY:
Preoperative Inclusion Criteria:

* Age ≥ 70 years
* Geriatric patients with hip fractures Treated either with oOsteosynthesis or oEndoprosthesis
* Ability of the patient or assigned representative to understand the content of the patient information / Informed Consent Form
* Signed and dated Institutional Review Board (IRB) / Ethics Committee (EC)-approved written informed consent

Preoperative Exclusion Criteria:

* Recent history of substance abuse (ie, recreational drugs, alcohol) that would preclude reliable assessment
* Prisoner
* Participation in any other medical device or medicinal product study within the previous month that could influence the results of the present study

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Primary care clinic (Usual Care clinic) Geriatric center
Sampling Method: Non-Probability Sample
Enrollment: 282 (Actual)
Dates: Start 2015-05; Primary Completion 2019-12 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
Major Adverse Events related to treatment / residential status / immobilization | From surgery up to 1 year follow-up
  Major AEs related to treatment / residential status / immobilization:
  * Delirium
  * Congestive heart failure
  * Pneumonia
  * Deep venous thrombosis
  * Pulmonary embolism
  * Pressure ulcers
  * Myocardial infarction

SECONDARY OUTCOMES:
Any other AEs not mentioned under primary outcome measure(s) as well as its relationship to the treatment / residential status / immobilization | From surgery up to 1 year follow-up
Activities of daily living | Baseline, 12 weeks and 1 year postoperative
  Modified Barthel index pre-injury, at 12 weeks and 12 months
Number of re-admissions to an acute hospital | From surgery up to 1 year follow-up
Timed up and go test (TUG) | 12 weeks and 1 year follow-up
Parker Mobility Score | Baseline, 12 weeks and 1 year follow-up
  Parker Mobility Score pre-injury, at 12 weeks and 12 months
Mortality | From surgery up to 1 year follow-up
Quality of Life | 12 weeks and 1 year postoperative
  Quality of life using the EuroQoL questionnaire (EQ-5D)
Pain | From surgery up to1 year follow-up
  Pain using the numeric rating scale
Direct and indirect costs | Baseline up to 1 year follow-up
  All direct and indirect costs will be documented for a cost-effectiveness analysis (medication, treatment, physiotherapy, postoperative care etc)
Time from admission to start of pain medication | Baseline (admission to surgery), about 1-2 days
Time from admission to start of fluid management | Baseline (admission to surgery), about 1-2 days
Time from admission to surgery | Baseline (admission to surgery), about 1-2 days
Time from surgery to discharge 1 and 2 | Baseline (admission to discharge), about 1-2 weeks
  Discharge 1 is defined as discharge from orthopaedic / trauma department Discharge 2 is defined as the timepoint when the patient is discharged to their definite residential status, i.e. residential status where no further change in residential status is planned . Discharge 1 and 2 may occur on the same date.
Residential status | Baseline up to 1 year follow-up
  Pre-injury, at discharge 1 and 2, at 12 weeks and 12 months
Falls | From surgery up to 1 year follow-up
  Numbers of falls
Medication | Baseline up to 1 year follow-up
  Number of different types of medication at admission, discharge 1, 12 weeks, 12 months and information whether analgesics, osteoporosis and other medications are administered at all study visit time points
Number of patients receiving adequate secondary fracture prevention | Baseline up to 1 year follow-up
Number of patients for which the nutrition status was evaluated / adapted | Baseline (admission to discharge), about 1-2 days
Occurrence of a contralateral hip fracture | Retrospective assessment of pre-injury status up to 1 year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Michael Blauth, Professor, Principal Investigator — Medical University of Innsbruck
Locations (12):
- United States (2):
  - Saint Louis University, St Louis, Missouri
  - Elmhurst Medical Center, New York, New York
- Austria (2):
  - Medical University of Innsbruck, Innsbruck
  - AKH Linz, Linz
- Netherlands (2):
  - Ziekenhuisgroep Twente, Almelo
  - Maastricht University Medical Center, Maastricht
- Singapore (2):
  - General Hospital Singapore, Singapore
  - Tan Tock Seng Hospital, Singapore
- Spain (2):
  - Hospital Son LLatzer, Palma de Mallorca, Balearic Island
  - Hospital Universitario Costa del Sol, Marbella
- Thailand (2):
  - Bhumibol Adulyadej Hospital, Bangkok
  - Hospital Medical Center Bangkok, Bangkok

REFERENCES:
- [Derived] Joeris A, Sprague S, Blauth M, Gosch M, Wattanapanom P, Jarayabhand R, Poeze M, Wong MK, Kwek EBK, Hegeman JH, Perez-Uribarri C, Guerado E, Revak TJ, Zohner S, Joseph D, Phillips MR. Cost-effectiveness analysis of the Geriatric Fracture Center (GFC) concept: a prospective multicentre cohort study. BMJ Open. 2023 Nov 2;13(11):e072744. doi: 10.1136/bmjopen-2023-072744. PMID 37918921
- [Derived] Blauth M, Joeris A, Rometsch E, Espinoza-Rebmann K, Wattanapanom P, Jarayabhand R, Poeze M, Wong MK, Kwek EBK, Hegeman JH, Perez-Uribarri C, Guerado E, Revak TJ, Zohner S, Joseph D, Gosch M. Geriatric fracture centre vs usual care after proximal femur fracture in older patients: what are the benefits? Results of a large international prospective multicentre study. BMJ Open. 2021 May 10;11(5):e039960. doi: 10.1136/bmjopen-2020-039960. PMID 33972329
- [Derived] Hurtado-Chong A, Joeris A, Hess D, Blauth M. Improving site selection in clinical studies: a standardised, objective, multistep method and first experience results. BMJ Open. 2017 Jul 12;7(7):e014796. doi: 10.1136/bmjopen-2016-014796. PMID 28706090
- [Derived] Joeris A, Hurtado-Chong A, Hess D, Kalampoki V, Blauth M. Evaluation of the geriatric co-management for patients with fragility fractures of the proximal femur (Geriatric Fracture Centre (GFC) concept): protocol for a prospective multicentre cohort study. BMJ Open. 2017 Jul 12;7(7):e014795. doi: 10.1136/bmjopen-2016-014795. PMID 28706089